CLINICAL TRIAL: NCT03422458
Title: The Impact of Immediate Implant Placement on Alveolar Ridge Preservation Techniques: a Clinical, Volumetric and Radiological Randomized Controlled Clinical Trial.
Brief Title: The Impact of Immediate Implant Placement on Alveolar Ridge Preservation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Principal Investigator, Marco Clementini, Research fellow, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-034
Record Dates: First submitted 2018-01-05; First posted 2018-02-05 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Post-Extraction Socket; Immediate Implant Placement; Alveolar Ridge Preservation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- natural healing (No Intervention): no treatment and the coagulum within the socket is left open for spontaneous healing
- Alveolar Ridge Preservation (Experimental): A bone substitute material (BioOss Collagen) is placed within the bony envelope at least to the level of the palatal/ lingual bone plate. Subsequently, the soft tissue borders of the alveole is de-epithelialized using a diamond drill under copious irrigation with water. A collagen matrix (Mucograft Seal) is adapted to the soft tissue borders again using single interrupted sutures.
  Interventions: Device: Alveolar Ridge Preservation
- Immediate Implant + Alveolar Ridge Preservation (Experimental): An immediate implant (Winsix) placement is performed. After implant insertion, a bone substitute material (BioOss Collagen) is placed in the gap occurred between the implant surface and the hard tissue walls of the extraction socket at least to the level of the palatal/ lingual bone plate. Subsequently, the soft tissue borders of the alveole is de-epithelialized using a diamond drill under copious irrigation with water. A collagen matrix (Mugograft Seal) is adapted to the soft tissue borders again using single interrupted sutures.
  Interventions: Device: Alveolar Ridge Preservation

INTERVENTIONS:
Device: Alveolar Ridge Preservation — Insertion of a bone substitute material (BioOss Collagen) within the bony envelope at least to the level of the palatal/ lingual bone plate. Adaptation of a collagen matrix (Mucograft Seal) to the soft tissue borders.
  Arms: Alveolar Ridge Preservation; Immediate Implant + Alveolar Ridge Preservation

SUMMARY:
It is well known that following the loss of a single tooth, severe hard- and soft-tissue alterations may take place within the affected site, resulting in a subsequent reduction of both vertical and horizontal ridge dimensions, often not allowing neither appropiate pontic fabrication nor correct placement of endosseous implants.

Over the past 20 years, various surgical procedures, grouped under the term of "alveolar ridge preservation" (ARP), have been introduced, aiming to maintain the existing soft and hard tissue envelope as well as a stable ridge volume, simplifying subsequent treatment procedures and optimizing functional and esthetic outcomes. They have been widely tested in controlled and not controlled clinical studies with various materials and approaches, and a number of recently published systematic reviews on this topic have confirmed the efficacy of ARP in preventing post-extraction dimensional changes of alveolar ridges.

After these procedures a minimum of four to six months must be awaited before implant insertion can be performed, bringing the patient compromised comfort, function and aesthetics and needing of a second surgical procedure for the implant placement.

Dental implant insertion at the time of tooth extraction (type I or immediate placement) reduced the number of dental appointments, of surgeries required and the overall treatment time. Nevertheless this surgical protocol does not provide predictable outcomes, since it may contribute towards a more pronounced bone resorption during healing. Different anatomical factors, as the thickness of the buccal bone wall and the dimension of the horizontal gap, may influence the dimensional changes of the alveolar crest following immediate implant placement. Such morphological changes could lead to negative esthetic complications, such as marginal soft tissues recessions, especially when affecting the buccal side of maxillary sites in patients with a high smile line.

It is unknown if immediate implant placement plus grafting materials and/or barrier membranes could influence post-extraction dimensional changes of alveolar ridges. No consensus exists on the need for bone augmentation simultaneously with immediate implant placement. Furthermore, no human study has yet compared dimensional changes of both hard and soft tissues after two different treatments: an alveolar ridge preservation technique for a subsequent implant placement, and an alveolar ridge preservation technique with an immediate implant placement.

DETAILED DESCRIPTION:
Hypothesis/Aims

Primary hypotesis

Placing an immediate implant into a fresh extraction site plus a bone substitute filling and a matrix covering could negatively modify the healing patterns and thus the tissue morphology of the ridge site with regard to:

* clinical hard tissues dimensions (bone width and height, bone volume)
* clinical soft tissues dimensions (soft tissues volume, keratinized tissues width and thickness, muco-gingival junction position's modifications, gingival color and texture,)

Secondary hypothesis.

Placing an immediate implant into fresh extraction site plus a bone substitute filling and a matrix covering could negatively influence tissue morphology of the preserved site with regard to:

* clinical hard tissues dimensions (bone width and height, bone volume)
* clinical soft tissues dimensions (soft tissues volume, keratinized tissues width and thickness, muco-gingival junction position's modifications, gingival color and texture,)

Aims:

The first aim of this study is to evaluate the possible impact on hard and soft tissue morphological changes of placing an immediate implant in post-extraction site treated by a bone substitute filling and a matrix covering.

The second aim of this study is to compare hard and soft tissue morphological changes in a spontaneous healed extraction site versus a fresh extraction site treated by immediate implant placement plus a bone substitute filling and a matrix covering

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years old) requiring extraction (for caries, fracture, periodontitis, prosthetic reasons) and subsequent moderately rough implant-supported single crown of one upper or lower asymptomatic front tooth or premolar
* Systemically healthy patients not smoking more than 10 cigarettes/day.
* Oral healty patients with adequate oral hygiene (bleeding on probing < 30%; Plaque index< 30%).

Exclusion Criteria:

* Patients smoking more than 10 cigarettes per day.
* Patients with oral mucosa diseases
* Patients with insulin-dependent diabetes.
* Patients with a history of malignancy, radiotherapy, or chemotherapy for malignancy.
* Patient pregnant or intended to be pregnant or nursing
* Patients taking medications or having treatments with an effect on mucosal healing in general (e.g. steroids, large doses of antiinflammatory drugs).
* Patients with a disease affecting connective tissue metabolism.
* Patients allergic to collagen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Hard tissue volumetric changes | 4 months
  Bone volumes changes at tooth extraction site
Soft tissue volumetric changes | 4 months
  Soft tissue volumes changes at tooth extraction site

SECONDARY OUTCOMES:
Keratinezed tissue (KT) | 4 months
  KT width changes at tooth extraction site

CONTACTS AND LOCATIONS:
Locations (1):
- Università Vita-Salute San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Derived] Clementini M, Castelluzzo W, Ciaravino V, Agostinelli A, Vignoletti F, Ambrosi A, De Sanctis M. The effect of immediate implant placement on alveolar ridge preservation compared to spontaneous healing after tooth extraction: Soft tissue findings from a randomized controlled clinical trial. J Clin Periodontol. 2020 Dec;47(12):1536-1546. doi: 10.1111/jcpe.13369. Epub 2020 Oct 21. PMID 32956551
- [Derived] Clementini M, Agostinelli A, Castelluzzo W, Cugnata F, Vignoletti F, De Sanctis M. The effect of immediate implant placement on alveolar ridge preservation compared to spontaneous healing after tooth extraction: Radiographic results of a randomized controlled clinical trial. J Clin Periodontol. 2019 Jul;46(7):776-786. doi: 10.1111/jcpe.13125. Epub 2019 May 31. PMID 31050359